CLINICAL TRIAL: NCT02728362
Title: Suprapatellar Nailing of Tibial Shaft Fractures: Long Term Follow Up
Brief Title: Suprapatellar Nailing of Tibial Shaft Fractures
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-027
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Broken Leg
Keywords: tibial shaft fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the functional outcomes and prevalence and severity of knee pain for patients undergoing suprapatellar nailing of tibial shaft fractures.

DETAILED DESCRIPTION:
Suprapatellar nailing...

Participants will be followed for 10 years prospectively. Follow up visits will occur at 2 weeks, 6weeks, 3 months, 6 months, 12 months, 3 years, 5 years, 7 years and 10 years.

Interim analysis will be done at 1, 3, 5, and 7 years with final analysis occuring at 10 years.

Primary and secondary endpoints in patients undergoing suprapatellar nailing of tibial shaft fractures are:

1. To evaluate the long term presence of knee pain
2. To evaluate the long term functional outcomes

ELIGIBILITY:
Inclusion Criteria:

* Isolated, unilateral tibial shaft fractures
* Orthopaedic Trauma Association (OTA) classification of 42 and may extend to 43A or 43B
* age 18-65, including pregnant women
* open or closed fractures
* able to sign consent
* english speaking

Exclusion Criteria:

* compartment syndrome
* other lower extremity injuries that will affect functional outcomes
* problems maintaining follow up (homeless, not willing to return for follow up)
* pathological fractures
* prisoners
* previous retained hardware in the injured leg
* injuries requiring vascular repair

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with tibial shaft fractures.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Long term presence of knee pain | 10 years
  During follow up visits participants will be administered the Visual Analog Scale (VAS) and the Patient Reported Outcomes Measurement Information System (PROMIS) Pain intensity short form 3a and Pain interference short form 8a. These forms will be analyzed together to determine an overall presence of knee pain.

SECONDARY OUTCOMES:
Long term functional outcomes | 10 years
  During follow up visits participants will be administered the Lysholm knee score and the PROMIS Mobility measure. These forms will be analyzed together to determine the overall long term function of the participants.
Knee Range of Motion (ROM) | 10 years
  During follow up visits the participants knee ROM will be measured
Fracture Healing | 10 years
  During follow up visits fracture healing will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Blake W Miller, DO, Principal Investigator — Corewell Health West

IPD SHARING:
Plan to Share IPD: No